CLINICAL TRIAL: NCT01461863
Title: Effects of Protein-calorie Supplementation on HIV Disease in Breastfeeding Women
Brief Title: DarDar Nutrition Study in HIV Breastfeeding Women
Acronym: DarDar2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, C. Fordham von Reyn, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD057614-03 (NIH); R01HD057614 (NIH)
Record Dates: First submitted 2011-10-13; First posted 2011-10-28 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Low Birth Weight
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protein calorie supplement (Active Comparator): 250 gm daily of specially designed porridge plus standard multivitamin
  Interventions: Dietary Supplement: Porridge protein calorie supplement
- Multivitamin (Placebo Comparator): Standard multivitamin control
  Interventions: Dietary Supplement: multivitamin

INTERVENTIONS:
Dietary Supplement: Porridge protein calorie supplement — 250 gm of fortified flour to make porridge containing 1062 kcal and 42 gm protein
  Other Names: Dar-uji
  Arms: protein calorie supplement
Dietary Supplement: multivitamin — Standard multivitamin
  Other Names: Darvite
  Arms: Multivitamin

SUMMARY:
This study being conducted in Dar es Salaam, Tanzania, to determine if a protein-calorie supplementation (PCS) and micronutrient supplement (MNS) will have an impact on health outcomes for HIV-infected pregnant women and their infants.

DETAILED DESCRIPTION:
In resource poor regions of the world where HIV is endemic, especially countries in sub-Saharan Africa, nutrition plays a critical role in HIV disease. Nutrition affects the health of HIV-infected women and children, and may influence the risk of mother to infant transmission of HIV through breast milk. Nutrition influences the risk of tuberculosis (TB) and TB disease severity. Existing research has focused on the role of micronutrients in HIV disease outcomes but has not addressed the role of protein calorie supplementation (PCS) in subpopulations of patients with HIV disease at high risk, specifically, HIV-infected women who are either breast feeding or have active TB. Our hypotheses are that administration of a culturally acceptable PCS is a practical, sustainable and effective strategy to: 1) decrease HIV viral load in plasma and breast milk of breast feeding women, enhance passively transferred immune mediators in breast milk, and improve HIV outcomes in women and their breast-fed infants and, 2) decrease HIV viral load, enhance TB-specific T cell immunity, and improve outcomes in women with HIV and active TB.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ women
* 2nd trimester of pregnancy
* Residency in Dar for duration of breastfeeding
* Plan to exclusively breastfeed

Exclusion Criteria:

* High risk pregnancy (e.g., diabetes, pre-eclampsia)
* Women with allergy to components of PCS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Fordham von Reyn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Magohe A, Mackenzie T, Kimario J, Lukmanji Z, Hendricks K, Koethe J, Neke NM, Tvaroha S, Connor R, Waddell R, Maro I, Matee M, Pallangyo K, Bakari M, von Reyn CF; DarDar-2 Study Team. Pre- and post-natal macronutrient supplementation for HIV-positive women in Tanzania: Effects on infant birth weight and HIV transmission. PLoS One. 2018 Oct 11;13(10):e0201038. doi: 10.1371/journal.pone.0201038. eCollection 2018. PMID 30307945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from HIV clinics in Dar es Salaam
Pre-assignment Details: Eligibility required that the woman be free of acute illness, have a BMI ≥18.5 kg/m2 and intend to exclusively breastfeed her infant for at least 3 months.
Period: Overall Study
Arm/Group | Protein Calorie Supplement | Multivitamin
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protein Calorie Supplement | Multivitamin | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 48 | 48 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 48 | 48 | 96
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Infant Weight
Description: Infant weight at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Protein Calorie Supplement | Multivitamin
Number analyzed (Participants) | 39 | 35
kg | 6.92 (0.82) | 7.32 (1.32)

2. Secondary Outcome: Maternal BMI at 9 Months
Description: Maternal BMI at 9 months
Time Frame: 9 months
Measure: Median (Standard Error); unit: kg/m^2
Groups:
- Multivitamin: Multivitamin
Arm/Group | Multivitamin | Protein Calorie Supplement
Number analyzed (Participants) | 36 | 41
kg/m^2 | 24.3 (1.1) | 23.8 (1.1)

ADVERSE EVENTS:
Arm/Group | Protein Calorie Supplement | Multivitamin
All-Cause Mortality (participants affected / at risk) | 1/48 | 1/48
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/48
Other Adverse Events (participants affected / at risk) | 0/48 | 4/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protein Calorie Supplement (N=48) | Multivitamin (N=48)
Death (Infections and infestations) | 1 (1) | 1 (1) — HIV infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protein Calorie Supplement (N=48) | Multivitamin (N=48)
Infant HIV infection (Infections and infestations) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes